CLINICAL TRIAL: NCT02892019
Title: A Multicenter, Randomized, Double-blind, Active-controlled, 2 Week Treatment, Parallel-group Study to Assess the Efficacy and Safety of Indacaterol Acetate Delivered Via the Concept1 Inhalation Device in Children Greater or Equal to 6 and Less Than 12 Years of Age With Asthma
Brief Title: Efficacy and Safety of Indacaterol Acetate Delivered Via the Concept1 Inhalation Device in Children Greater or Equal to 6 and Less Than 12 Years of Age With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQMF149G2202; 2016-002113-21 (EudraCT Number)
Record Dates: First submitted 2016-09-01; First posted 2016-09-08 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Asthma
Keywords: indacaterol acetate, asthma, GINA 2015, pediatrics
MeSH Terms: conditions — Asthma | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indacaterol acetate 75 μg o.d. (Active Comparator): Indacaterol acetate 75 μg o.d. delivered via Concept1 inhaler
  Interventions: Drug: Indacaterol acetate 75 μg
- Indacaterol acetate 150 μg o.d. (Active Comparator): Indacaterol acetate 150 μg o.d. delivered via Concept1 inhaler
  Interventions: Drug: Indacaterol acetate 150 μg

INTERVENTIONS:
Drug: Indacaterol acetate 75 μg — Indacaterol acetate 75 μg o.d. delivered via Concept1 inhaler
  Other Names: QAB149
  Arms: Indacaterol acetate 75 μg o.d.
Drug: Indacaterol acetate 150 μg — Indacaterol acetate 150 μg o.d. delivered via Concept1 inhaler
  Other Names: QAB149
  Arms: Indacaterol acetate 150 μg o.d.

SUMMARY:
This study is designed to explore lung function effects of two doses of indacaterol acetate, 75 μg and 150 μg, in pediatric asthma patients 6-11 years old, and to compare the systemic exposure to indacaterol in plasma with historical data in adults, to identify an appropriate dose to Phase III evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children ≥ 6 years and < 12 years with confirmed diagnosis of asthma for at least 1 year prior to study enrollment.
* Written informed consent by parent(s)/legal guardian(s) and depending upon their age and local requirements a consent or assent for the patient.
* Patients receiving daily treatment with a stable low dose Inhaled Corticosteroid (ICS) (with or without additional controller), or patients receiving daily treatment with a stable mid-dose ICS (monotherapy or together with LTRA) for at least 4 weeks prior to Screening, and able to tolerate fluticasone propionate 100 μg b.i.d. inhaler starting at Visit 1 (or soon after).
* Patients with a pre-bronchodilator FEV1 ≥ 50% and ≤ 90% of the predicted normal value for the patient at the start and end of Run-in (Visits 101 and 199).
* Patients who demonstrate an increase in FEV1 of 12% within 30 minutes after administration of 400 μg salbutamol/360 μg albuterol (or equivalent dose) at Visit 101. All patients must perform a reversibility test at Visit 101.

Exclusion Criteria:

* Patients taking a mid-dose ICS (per GINA guidelines) in combination with LABA or any patient taking high-dose ICS.
* Evidence of unstable disease within 4 weeks prior to Screening (Visit 1).
* Patients who have had an asthma attack/exacerbation requiring systemic steroids (SCS) or hospitalization or emergency room visit within 3 months prior to Visit 1 (Screening) or more than 3 separate exacerbations in the 12 months preceding Visit 1.
* Suspected or documented bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear that is not resolved within 4 weeks of Screening (Visit 1).
* Prior intubation for asthma.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (26):
- Belgium (2):
  - Novartis Investigative Site, Bruges
  - Novartis Investigative Site, Brussels
- Colombia (2):
  - Novartis Investigative Site, Bogotá
  - Novartis Investigative Site, Bucaramanga
- Croatia (2):
  - Novartis Investigative Site, Slavonski Brod
  - Novartis Investigative Site, Zagreb
- Germany (3):
  - Novartis Investigative Site, Hamm
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Rosenheim
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, GTM
  - Novartis Investigative Site, Guatemala City
- Hungary (4):
  - Novartis Investigative Site, Törökbálint, Pest County
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
  - Novartis Investigative Site, Szigetvár
- Philippines (3):
  - Novartis Investigative Site, Manila, National Capital Region
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Novartis Investigative Site, Saint Petersburg, Russia
- Slovakia (2):
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Nové Zámky, SVK
- South Africa (3):
  - Novartis Investigative Site, Middelburg, Mpumalanga
  - Novartis Investigative Site, Panorama, Western Cape
  - Novartis Investigative Site, Cape Town
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Sekerel BE, Nell H, Laki I, Pak T, Contreras E, Kolarz A, D'Andrea P, Manga V, Jain M, Vaidya S, Valentin M, Sen B. Efficacy, Safety, and Systemic Exposure of Once-Daily Indacaterol Acetate in Pediatric Asthma: A Randomized, Double-Blind, Controlled Dose-Finding Study. Clin Drug Investig. 2023 Sep;43(9):719-728. doi: 10.1007/s40261-023-01300-8. Epub 2023 Sep 8. PMID 37682405

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: randomized set : 80 participants (41 and 39) Full analysis set : 79 participants (41 and 38) safety set : 79 participants (41 and 38) per protocol set : 35 participants (35 and 34)
Period: Overall Study
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Started | 41 | 39
Completed | 40 | 36
Not Completed | 1 | 3
Not completed — randomized but not treated | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d. | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.3 (1.47) | 9.1 (1.58) | 9.2 (1.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 28 | 24 | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 17 | 17 | 34
  Black | 3 | 3 | 6
  Asian | 1 | 3 | 4
  Native American | 3 | 3 | 6
  Unknown | 1 | 0 | 1
  Other | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratoty Volume in 1 Second (FEV1)
Description: Change from baseline in pre-dose trough FEV1 after 2 weeks of treatment with indacaterol acetate 75 μg o.d and 150 μg o.d.
  The primary endpoint is change from baseline in pre-dose trough FEV1 (mL) after 2 weeks of treatment. The pre-dose trough FEV1 (mL) is defined as the mean of the two FEV1 (mL), values measured at -45 min and -15 min pre-dose.
Time Frame: 2 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Number analyzed (Participants) | 41 | 38
L | 0.171 (0.1664) | 0.212 (0.2521)

2. Secondary Outcome: Systemic Exposure to Indacaterol in Plasma
Description: Systemic exposure to indacaterol in plasma following sparse pharmacokinetic (PK) sampling on Day 1 and Day 14 after inhalation of indacaterol acetate 75 μg and 150 μg.
Time Frame: day 1, day 14
Population: safety set
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Number analyzed (Participants) | 41 | 38
pg/mL
  Day 1 <=-2 hours: number analyzed (Participants) | 35 | 31
  Day 1 <=-2 hours | 0.0 (0.0) | 0.0 (0.0)
  Day 1, 15 minutes: number analyzed (Participants) | 37 | 34
  Day 1, 15 minutes | 204.1 (98.27) | 73.7 (39.55)
  Day 1, 1 hour: number analyzed (Participants) | 36 | 32
  Day 1, 1 hour | 125.8 (63.13) | 43.9 (20.84)
  Day 14 <=-2 hours: number analyzed (Participants) | 38 | 31
  Day 14 <=-2 hours | 80.9 (32.51) | 46.7 (29.61)
  Day 14, 15 minutes: number analyzed (Participants) | 41 | 35
  Day 14, 15 minutes | 393.1 (182.11) | 137.3 (47.43)
  Day 14, 1 hour: number analyzed (Participants) | 41 | 34
  Day 14, 1 hour | 255.5 (117.67) | 103.0 (37.88)

3. Secondary Outcome: Asthma Control as Assessed by Pediatric Interviewer-administered Asthma Control Questionnaire
Description: Asthma Control as assessed by pediatric interviewer-administered Asthma Control Questionnaire (ACQ-IA) score at week 2 (mean change). A decrease in the score shows an improvement.
  The scale ranges from 0 (no symptoms) to 6 (severe symptoms every day). Results are given as a change as compared from baseline
Time Frame: 2 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Number analyzed (Participants) | 41 | 38
score on a scale | -0.375 (0.3796) | -0.270 (0.6341)

4. Secondary Outcome: Pre-dose Morning and Evening Peak Expiratoty Flow (PEF)
Description: Pre-dose morning and evening PEF over 2 weeks of treatment as determined by electronic peak flow meter data (mean change)
Time Frame: 2 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Number analyzed (Participants) | 41 | 38
L/min
  Morning PEF: number analyzed (Participants) | 39 | 37
  Morning PEF | 29.6 (26.41) | 14.7 (29.38)
  Evening PEF: number analyzed (Participants) | 39 | 37
  Evening PEF | 29.7 (25.57) | 15.2 (28.58)

5. Secondary Outcome: Rescue Medication Usage (Mean Daiily Number of Puffs)
Description: Rescue medication usage over 2 weeks of treatment as determined by patient diary data for indacaterol acetate 75 μg and 150 μg o.d.Results given as mean change of puffs of rescue medication.
Time Frame: 2 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: number of puffs
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Number analyzed (Participants) | 41 | 38
number of puffs | -0.19 (1.479) | -0.22 (0.930)

6. Secondary Outcome: Rescue Medication Usage (Percentage of Rescue Medication Free Days)
Description: Rescue medication usage over 2 weeks of treatment as determined by patient diary data for indacaterol acetate 75 μg and 150 μg o.d.
Time Frame: 2 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Number analyzed (Participants) | 41 | 38
percentage | 7.4 (22.37) | 3.1 (19.42)

7. Secondary Outcome: Forced Expiratoty Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC)
Description: FEV1 and FVC at 30 minutes and 1-hour post dose at week 2 for indacaterol acetate 75 μg and 150 μg o.d.
Time Frame: 2 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Number analyzed (Participants) | 41 | 38
L
  30 minutes: number analyzed (Participants) | 40 | 34
  30 minutes | 0.234 (0.1786) | 0.224 (0.2459)
  1 hour: number analyzed (Participants) | 40 | 35
  1 hour | 0.224 (0.1725) | 0.258 (0.2451)

8. Secondary Outcome: Symptoms as Recorded by Patient E-diary (Mean Total Daily Symptom Score)
Description: Symptoms as recorded by patient e-diary for indacaterol acetate 75 μg and 150 μg o.d. (mean change) The scale rages from 0 (no problem) - 4 (very severe problems).
Time Frame: 2 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Number analyzed (Participants) | 41 | 38
score on a scale | -0.18 (0.695) | 0.08 (0.365)

9. Secondary Outcome: Symptoms as Recorded by Patient E-diary (Percentage of Asthma Symptoms Free Days)
Description: Symptoms as recorded by patient e-diary for indacaterol acetate 75 μg and 150 μg o.d. (mean change)
Time Frame: 2 weeks
Population: full analysis set
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Indacaterol Acetate 150 μg o.d. | Indacaterol Acetate 75 μg o.d.
Number analyzed (Participants) | 41 | 38
percentage | 12.3 (21.25) | 4.4 (26.60)

ADVERSE EVENTS:
Time Frame: 2 years
Description: AE additional description
Groups:
- QAB149 150 ug OD: QAB149 150 ug OD
- QAB149 75 ug OD: QAB149 75 ug OD
Arm/Group | QAB149 150 ug OD | QAB149 75 ug OD
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/38
Other Adverse Events (participants affected / at risk) | 3/41 | 13/38
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QAB149 150 ug OD (N=41) | QAB149 75 ug OD (N=38)
Defect conduction intraventricular (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Peak expiratory flow rate decreased (Investigations) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT02892019/SAP_000.pdf
  • Study Protocol (2016-06-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT02892019/Prot_001.pdf